CLINICAL TRIAL: NCT01540708
Title: An Open-label, Randomised, Cross-over, Single Centre Study in Healthy Volunteers to Optimise the Rotacap Formulation andROTAHALER Device for Delivery of Fluticasone Propionate/Salmeterol.
Brief Title: A Single Centre Study in Healthy Volunteers to Optimise the Rotacap Formulation and ROTAHALER Device for Delivery of Fluticasone Propionate/Salmeterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116409
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Asthma; Respiratory; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SERETIDE Rotacaps (Experimental): Fluticasone propionate/Salmeterol combination administered at 2 doses (250/50 mcg and 100/50 mcg) and delivered in a capsule-based inhaler (Rotahaler). Devices with varying airflow resistance, low, intermediate and high, will be used.
  Interventions: Drug: SERETIDE Diskus
- SERETIDE Diskus (Active Comparator): Fluticasone propionate/Salmeterol combination administered at 2 doses (250/50 mcg and 100/50 mcg) and delivered in a multi-dose dry powder inhaler
  Interventions: Drug: SERETIDE Rotacaps

INTERVENTIONS:
Drug: SERETIDE Rotacaps — The study will be conducted in 3 parts with an adaptive design where pharmacokinetic data analysis follows each part to enable a decision on whether progression to the subsequent parts is required. Thirty six subjects will be enrolled in each part. Part A will test an alternative version of the Rotahaler with a lower airflow resistance. The study will then test one or more of the following options depending on the outcome of part A. If progressed, part B will test modified Rotacap formulations including: (1) modified blend formulation, (2) reduced capsule fill weights, (3) different capsule types. Part B will also test other versions of the Rotahaler with intermediate airflow resistance. Part C will test the lower strength FP/salmeterol (100/50 mcg or lower) and/or a new unit dose DPI device (BUDI). In each arm, subjects will be administered 7 doses (3.5 days bid) with PK sampling following administration of the 7th dose on the morning of Day 4.
  Arms: SERETIDE Diskus
Drug: SERETIDE Diskus — The study will be conducted in 3 parts with an adaptive design where pharmacokinetic data analysis follows each part to enable a decision on whether progression to the subsequent parts is required. Thirty six subjects will be enrolled in each part. Part A will test an alternative version of the Rotahaler with a lower airflow resistance. The study will then test one or more of the following options depending on the outcome of part A. If progressed, part B will test modified Rotacap formulations including: (1) modified blend formulation, (2) reduced capsule fill weights, (3) different capsule types. Part B will also test other versions of the Rotahaler with intermediate airflow resistance. Part C will test the lower strength FP/salmeterol (100/50 mcg or lower) and/or a new unit dose DPI device (BUDI). In each arm, subjects will be administered 7 doses (3.5 days bid) with PK sampling following administration of the 7th dose on the morning of Day 4.
  Arms: SERETIDE Rotacaps

SUMMARY:
The purpose of this study is to optimise the device and/or formulation of the Fluticasone propionate (FP)/salmeterol (SALM) unit dose powder inhaler (Rotahaler) to achieve drug delivery characteristics comparable to the Fluticasone propionate /salmeterol DISKUS inhaler. The indication is asthma and chronic obstructive pulmonary disease. The study is an open-label, randomised, cross-over, single centre study in healthy volunteers and will be conducted in a maximum of 3 parts, A, B and C. The design is adaptive and pharmacokinetic (PK) data analysis follows each part to enable a decision on whether progression to the subsequent parts is required.

Part A of the study will test an alternative version of the Rotahaler with a low airflow resistance. The study will then test one or more of the following options depending on the outcome of part A. If progressed, part B will test modified Rotacap formulations including: (1) modified blend formulation, (2) reduced capsule fill weights, (3) different capsule types. Part B will also test other versions of the Rotahaler with intermediate airflow resistance. Part C will test the lower strength FP/salmeterol (100/50 mcg or lower) and/or a new unit dose DPI device (BUDI).

A total of 36 subjects will be enrolled in each part to ensure 32 complete. In each cross-over arm, subjects will be administered 7 doses (3.5 days bid) with PK sampling following administration of the 7th dose. A three-day minimum wash-out period will separate each cross-over arm.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a chronic inflammatory disease of the airways characterised by varying and recurring symptoms of shortness of breath, chest tightness, wheezing and cough, airflow obstruction, bronchial hyper-responsiveness and underlying inflammation.

The GINA guidelines [Global Initiative for Asthma,(GINA) updated 2009] highlight the need to treat airway inflammation in asthma and recognise the importance of inhaled prophylactic medications such as inhaled corticosteroids and combinations of Inhaled Corticosteroids (ICS) / Long Acting Beta Agonists (LABA) such as SERETIDE™ for the treatment of chronic asthma.

Chronic obstructive pulmonary disease (COPD) is a preventable and treatable disease characterised by airflow limitation that is not fully reversible [Celli, 2004]. The airflow limitation of COPD is primarily due to small airways disease and parenchymal destruction associated with an abnormal inflammatory response of the lungs, mainly caused by cigarette smoking [Celli 2004]. COPD is characterised by symptoms of chronic and progressive breathlessness (or dyspnea), cough and sputum production which can be a major cause of disability and anxiety associated with the disease.

The GOLD (Global Strategy for the Diagnosis, Management and Prevention of Chronic Obstructive Pulmonary Disease) guidelines on COPD state that the goals of pharmacologic therapy should be to control symptoms, improve health status and exercise tolerance, and reduce the frequency of COPD exacerbations [GOLD, 2008]. Research has indicated that an inhaled corticosteroid (ICS) combined with a long acting β2-agonist (LABA) is more effective than the individual components in managing stable COPD to reduce exacerbations and improve lung function and health status [Ferguson, 2008; Calverley, 2007; Kardos, 2007].

The efficacy of the combination product, SERETIDE has been established in the metered dose inhaler (MDI) and multidose powder inhaler (Ddpi; DISKUS™/Accuhaler) in both asthma and Chronic Obstructive Pulmonary Disease, COPD at a variety of dose strengths.

Alternative treatment options with respect to the formulation of SERETIDE and its means of delivery via an inhaler device are currently being assessed by GSK with a view to developing a product with bioavailability characteristics comparable to those of SERETIDE delivered via the multi-dose powder inhaler (DISKUS™/Accuhaler). It is intended that the product will then be progressed for treatment administration in both asthma and COPD patients.

STUDY RATIONALE:

A recently completed study, ASR114334, [GlaxoSmithKline document number YM2010/00082/02] evaluated the comparative bioavailability of fluticasone propionate/salmeterol delivered via the established multi-dose powder inhaler (Ddpi, DISKUS/Accuhaler) with the Rotahaler unit dose fluticasone propionate/salmeterol capsule-based powder inhaler (Rdpi) in both asthma and COPD patients. The Rotahaler (Rdpi) inhaler had an airflow resistance similar to the DISKUS multi-dose inhaler (Ddpi). Whilst the active ingredients were a combination of fluticasone propionate/salmeterol, the devices were different with respect to their handling and instructions for operation, although both were designed to deliver at the 250/50mcg bid dose strength ie mcg equivalent doses.

The results showed that plasma exposures of both fluticasone propionate (FP) and salmeterol were 1.5 to 2 fold higher following repeat dose administration of FP/salmeterol delivered from the Rdpi compared with those from the Ddpi, [GlaxoSmithKline document number 2011N112456_00]. This was observed for both asthma and COPD patients.

The purpose of this study, ASR116409 is to optimise the device and/or formulation of the FP/salmeterol unit dose powder inhaler to achieve drug delivery characteristics comparable to the FP/salmeterol DISKUS.

DOSE RATIONALE:

Two doses of FP/salmeterol will be administered in this study: 250/50 mcg and 100/50 mcg or lower, both doses are approved for the treatment of asthma. These doses will be administered to healthy subjects and are at or below the maximum approved doses for FP and salmeterol indicated for chronic therapy in asthma; therefore there are no anticipated safety concerns associated with the planned short term (3.5 days bid) dosing in healthy subjects.

STUDY DESIGN:

The study is an open-label, randomised, cross-over, single centre study in healthy volunteers in 3 parts, A, B and C. It will be conducted with an adaptive design where pharmacokinetic data analysis follows each part to enable a decision on whether progression to the subsequent parts is required.

A total of 36 subjects will be enrolled in each part to ensure 32 complete. In each cross-over arm, subjects will be administered 7 doses (3.5 days bid) with PK sampling following administration of the 7th dose. A three-day minimum wash-out period will separate each cross-over arm. Subjects may elect to participate in more than one part.

Part A will compare the bioavailability characteristics of the following GSK devices: the Ddpi (multi-dose dry powder inhaler, DISKUS), the Rdpi(H) (capsule-based inhaler, high airflow resistance) and the Rdpi(L) (low airflow resistance). The Rdpi(H) has higher airflow resistance to the Ddpi compared to the Rdpi (L) and could allow a closer PK match. Part A will consist of a four treatment cross-over sub-study with the following arms, each arm replicated twice for each subject.

Treatment arms for part A will comprise:

* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Ddpi
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Rdpi(H). Instructions for subjects will be to take 2 steady, deep inhalations.
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Rdpi(L). Instructions for subjects will be to take 1 fast and deep inhalation
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Rdpi(L). Instructions for subjects will be to take fast and deep inhalations until no powder remains in the inhaler.

The Rdpi(H) device (250/50mcg FP/salmeterol) is being assessed in Part A to bridge the data back to the previous study (ASR114334) to show whether it is possible to replicate the 1.5 to 2 fold systemic exposure ratio for Rdpi(H)/Ddpi in healthy subjects compared to patients seen in the previous study (ASR114334).

Subjects will be dosed twice daily for 3 days and once on the fourth day in the morning. The first dose on Day 1 will be administered at the site and the next four doses will be self-administered by the subjects at home. They will attend the Unit in the evening of the 3rd day where they will be administered the 6th dose and remain at the Unit for the night and following day. They will be dosed in clinic (7th dose) on the morning of the fourth day and remain at site until completion of the 12 hour post-dose PK sample collection.

Following a 3-day minimum wash-out period after the last dose of study medication (Day 4), subjects will participate in the subsequent arms of Part A until they have completed all 4 arms twice i.e. the 8 periods planned for completion of Part A.

PK samples will be analysed and reviewed at the conclusion of Part A. If PK equivalence for FP and SALM is demonstrated between the Rdpi(L)and the Ddpi, and Rdpi(H)is demonstrated to have higher and non-equivalent PK systemic exposure compared to Ddpi, Part C will be conducted. If PK equivalence is not demonstrated, Part B will be conducted.

Part B: Study design for Part B will depend on the PK results from Part A. Prior to the start of part B, a decision will be made by the sponsor team as to whether the Rdpi (H) or the Rdpi(L) device will be used; this decision will be based on PK data from part A. FP/Salm 250/50mcg from the Ddpi will be included again in Part B as a control group.

If the plasma exposures of FP and SALM obtained during Part A from Rdpi(H) are statistically higher than those from the Dpi and those from Rdpi (L) are statistically lower than those from the Ddpi, Part B will assess two intermediate airflow resistance versions of the Rdpi [Rdpi (IM)] and/or the formulation changes below:

* modified blend formulations
* reduced capsule fill weights,
* different capsule types If the plasma exposures of FP and SALM obtained from the Rdpi(H) are statistically higher than those from the Dpi and those from the Rdpi(L) are statistically higher than those from the Ddpi, Part B will assess the formulation changes below using Rdpi(H);
* modified blend formulations
* reduced capsule fill weights,
* different capsule types One variable will be assessed at a time in an open-label, randomized, cross-over manner comprising 2 to 3 arms separated by a 3-day minimum wash-out period. All comparisons will be done against the DISKUS arm, in order to test bioequivalence. The sample size and the use of replicated arms will be evaluated and defined after the completion of part A, adapting the design and the sample size to the variability observed during the previous part of the study.

Following PK data analysis for all the variables, two or more variables may finally be grouped for combined assessment as an open-label investigation.

Evaluation of the two intermediate high airflow resistance Rdpi devices [Rdpi(IM)] and of the formulation changes will be conducted in a cross-over design. The inhalation instructions (number and type of breaths) will be decided after Part A is completed. An additional arm whereby subjects will be administered the Ddpi will also be included for comparison.

Part C will compare bioavailability parameters for 2 dosage strengths of FP/salmeterol: 100/50 mcg, and 250/50mcg, delivered from the Ddpi and the device/formulation shown to demonstrate bioequivalence in Part A and/or Part B.

Another GSK unit dose device in development, the BUDI inhaler, will also be evaluated for its comparative bioavailability characteristics at both doses.

If PK data from Part A demonstrates that the Rdpi(L) is PK equivalent to the Ddpi at the 250/50 mcg dose, Part B will not be conducted. We will also test the bovine capsule which may be needed for certain markets in Part C if Part B is not conducted.

The various arms in Part C will not be conducted concurrently as timing of dosing for each arm will depend on availability of study medication, device and capsule type.

Part C will therefore be conducted at two different points in time: Part C1 will consist of a 3 or 4-way cross-over sub-study with the following arms:

* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Ddpi
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (100/50mcg) delivered via the Ddpi
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (100/50mcg) delivered via the device/formulation combination selected in Part A or B
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Bovine capsule (if part B is not performed).

Part C2 will be performed if required when the BUDI inhaler will be made available, a cross-over sub-study with the following arms:

* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via the Ddpi
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (100/50mcg) delivered via the Ddpi
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (250/50mcg) delivered via BUDI Inhaler
* Administration of 7 doses (3.5 days bid) of FP/salmeterol (100/50mcg) delivered via the BUDI Inhaler.

The inhalation instructions (number and type of breaths) will be decided after part A is completed

The option to combine Parts C1 and C2 will be evaluated according to the:

* availability of the BUDI Inhaler and the timing of Part C
* PK results from the previous parts (variability could affect the need to have replicated arms in part C as well; further, the bovine capsule may have been already tested in part B).

PRIMARY OBJECTIVES:

* To select a device and formulation combination of fluticasone propionate/salmeterol (250/50mcg or lower) which has pharmacokinetic equivalence (ratio 0.8 to 1.25) to fluticasone propionate/salmeterol (250/50mcg) delivered via the Ddpi (multi dose dry powder inhaler)
* To compare the pharmacokinetic parameters of fluticasone propionate/salmeterol (250/50mcg or lower) delivered from a range of devices and/or formulations to those of fluticasone propionate/salmeterol (250/50mcg) delivered via the Ddpi in healthy volunteers.

SECONDARY OBJECTIVES:

* To determine the pharmacokinetic equivalence of the selected device/formulation combination of fluticasone propionate/salmeterol administered at a lower dose to match fluticasone propionate/salmeterol administered at the 100/50mcg dose from the Ddpi
* To assess the PK characteristics of the BUDI inhaler containing 100/50mcg fluticasone propionate/salmeterol and 250/50mcg fluticasone propionate/salmeterol.

PRIMARY ENDPOINT:

-Pharmacokinetic endpoint: Area under the plasma fluticasone propionate concentration-time curve over dosing interval ; maximum observed concentration for fluticasone propionate and salmeterol plasma concentration-time curve on the last day of each study treatment period (Day 4).

SECONDARY ENDPOINT:

-Pharmacokinetic parameters: time of maximum observed concentration;terminal phase rate constant; terminal phase half-life for fluticasone propionate and salmeterol) on the last day of each treatment period (Day 4).

TREATMENT ASSIGNMENT:

During Part A of the study, subjects will be assigned to one of the four sequences of the below reported table (4x4 Williams design with replicates) in accordance with the randomization schedule generated by Quantitative Sciences, prior to the start of the study, using validated internal software.

Sequence number Arm

1. A B D C D A C B
2. B C A D C D B A
3. C D B A B C A D
4. D A C B A B D C

A indicates Ddpi, B indicates Rdpi(H), C indicates Rdpi(L) fast and deep inhalation, and D indicates Rdpi(L) fast and deep inhalations until no powder remains in the inhaler.

Williams design, with replicates or not, will be adopted for the subsequent and optional parts of the study, depending on the results obtained in part A.

ELIGIBILITY:
INCLUSION CRITERIA:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single QTc, QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the protocol approved contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential and is abstinent or agrees to use one of the protocol approved contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit
* Capable of giving informed consent, which includes compliance with the study requirements and restrictions listed in the consent form.
* BMI within the range 18 and 35 kg/m2 (inclusive).
* Able to use the inhaler devices adequately after training

EXCLUSION CRITERIA:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Medical Condition Exclusions:

* Subjects who have a current diagnosis or a history of asthma, excluding childhood asthma which has been discharged by physician (e.g., for any FTIH where risk of bronchoconstriction is unknown, or compound specific where risk of bronchoconstriction). This must be documented in the subject's medical notes.
* Subjects who have a current and previous diagnosis of COPD. This must be documented in the subject's medical notes.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Subject is mentally or legally incapacitated.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Medical Exclusions:

* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Lifestyle Exclusions:

* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the screening visit defined by the following Australian guidelines as:

Males: An average weekly intake greater than 21 units or an average daily intake greater than 3 units. Females: An average weekly intake greater than 14 units or an average daily intake greater than 2 units.

One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.

* Grapefruit, pummelos, or grapefruit juice containing products are excluded from 2 weeks prior to randomisation (all study parts) until collection of the final blood sample on Day 4.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2012-09-04 (Actual); Study Completion 2012-09-04 (Actual)

PRIMARY OUTCOMES:
Selection of a device and formulation combination of fluticasone propionate/salmeterol (250/50mcg or lower) which has pharmacokinetic equivalence (ratio 0.8 to 1.25) to fluticasone propionate/salmeterol (250/50mcg) delivered via the Ddpi | PK on Day 4 of each treatment arm: 0, 5, 10, 30 min and 1, 2, 4, 8, 10 and 12 hours post-dose
Comparison of he pharmacokinetic parameters of fluticasone propionate/salmeterol (250/50mcg or lower) delivered from a range of devices and/or formulations to those of fluticasone propionate/salmeterol (250/50mcg) delivered via the Ddpi | PK on Day 4 of each treatment arm: 0, 5, 10, 30 min and 1, 2, 4, 8, 10 and 12 hours post-dose
  Area under the plasma fluticasone propionate concentration-time curve over dosing interval; maximum concentration for fluticasone propionate and salmeterol plasma concentration-time curve on the last day of each study treatment period (Day 4).

SECONDARY OUTCOMES:
Determination of the pharmacokinetic equivalence of the selected device/formulation combination of fluticasone propionate/salmeterol administered at a lower dose to match fluticasone propionate/salmeterol administered at 100/50mcg dose from Ddpi | PK on Day 4 of each treatment arm: 0, 5, 10, 30 min and 1, 2, 4, 8, 10 and 12 hours post-dose
  Pharmacokinetic parameters: time of maximum observed concentration;terminal phase rate constant; terminal phase half-life for fluticasone propionate and salmeterol) on the last day of each treatment period (Day 4).
Assessment of the PK characteristics of the BUDI inhaler containing 100/50mcg fluticasone propionate/salmeterol and 250/50mcg fluticasone propionate/salmeterol | PK on Day 4 of each treatment arm: 0, 5, 10, 30 min and 1, 2, 4, 8, 10 and 12 hours post-dose
  Pharmacokinetic parameters: time of maximum observed concentration;terminal phase rate constant; terminal phase half-life for fluticasone propionate and salmeterol) on the last day of each treatment period (Day 4).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Yates JC, Vestbo J; TORCH investigators. Salmeterol and fluticasone propionate and survival in chronic obstructive pulmonary disease. N Engl J Med. 2007 Feb 22;356(8):775-89. doi: 10.1056/NEJMoa063070. PMID 17314337
- [Background] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Background] Ferguson GT, Anzueto A, Fei R, Emmett A, Knobil K, Kalberg C. Effect of fluticasone propionate/salmeterol (250/50 microg) or salmeterol (50 microg) on COPD exacerbations. Respir Med. 2008 Aug;102(8):1099-108. doi: 10.1016/j.rmed.2008.04.019. Epub 2008 Jul 9. PMID 18614347
- [Background] GINA: Global strategy for asthma management and prevention. NHLBI/WHO/GARD, Washingon DC 2006-updated 2009.
- [Background] GlaxoSmithKline Document Number RM2007/00413/03. CCI18781+GR33343 Investigator's Brochure, version number 12, dated 4 May 2011.
- [Background] GlaxoSmithKline document number YM2010/00082/02 Study ASR114334: A comparative bioavailability study to compare the pharmacokinetics and pharmacodynamic effects of Fluticasone propionate and Salmeterol delivered by Fluticasone propionate/ Salmeterol combination in a capsule-based inhaler and a multi-dose dry powder inhaler, in patients with moderate asthma and patients with moderate to severe COPD.
- [Background] GOLD 2006 Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease (2006)-updated 2009.
- [Background] James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, Davern TJ, Lee WM. Pharmacokinetics of acetaminophen-protein adducts in adults with acetaminophen overdose and acute liver failure. Drug Metab Dispos. 2009 Aug;37(8):1779-84. doi: 10.1124/dmd.108.026195. Epub 2009 May 13. PMID 19439490
- [Background] Kardos P, Wencker M, Glaab T, Vogelmeier C. Impact of salmeterol/fluticasone propionate versus salmeterol on exacerbations in severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Jan 15;175(2):144-9. doi: 10.1164/rccm.200602-244OC. Epub 2006 Oct 19. PMID 17053207
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Result] GlaxoSmithKline document number 2011N112456_00 Study report for A comparative bioavailability study to compare the pharmacokinetics and pharmacodynamic effects of fluticasone propionate and salmeterol delivered by fluticasone propionate/salmeterol combination in a capsule-based inhaler and a multi-dose dry powder inhaler, in patients with moderate asthma and patients with moderate to severe COPD.
- See also: Results for study 116409 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116409?search=study&search_terms=116409#rs